CLINICAL TRIAL: NCT02375867
Title: Safety and Efficacy of Steroids in the Management of Fulminant Hepatic Failure Due to Hepatitis A Virus in the Pediatric Age Group
Brief Title: Steroids in Fulminant Hepatitis A in the Pediatric Age Group
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Liver Institute, Egypt (Other)
Collaborators: Quesna Central Hospital, Ministry Of Health, Egypt (Unknown)
Responsible Party: Principal Investigator, Mostafa M. Sira, Associate Professor of Pediatric Hepatology, National Liver Institute, Egypt
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: NLI-FHF-S-PED
Record Dates: First submitted 2015-02-14; First posted 2015-03-03 (Estimated); Last update posted 2018-12-17 (Actual); Status verified 2018-12

CONDITIONS: Fulminant Hepatic Failure
MeSH Terms: conditions — Liver Failure, Acute | interventions — Prednisolone; Methylprednisolone; Methylprednisolone Hemisuccinate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- prednisolone (Active Comparator): This group includes patients with FHF without encephalopathy
  Interventions: Drug: prednisolone
- methylprednisolone (Active Comparator): This group includes patients with FHF with encephalopathy
  Interventions: Drug: methylprednisolone
- Non-intervention (No Intervention): FHF patients without any of the proposed intervention as controls

INTERVENTIONS:
Drug: prednisolone — Oral administration of 1 mg/Kg/day
  Other Names: Hostacortin-H
  Arms: prednisolone
Drug: methylprednisolone — Intravenous injection of 0.8 mg/kg/day
  Other Names: Solumedrol
  Arms: methylprednisolone

SUMMARY:
Fulminant hepatic failure (FHF) in children is a potentially devastating disease. The mortality rate may reach 80-90% in the absence of liver transplantation. Liver injury is considered to be mainly immune mediated with augmentation of cytolytic pathways of infected hepatocytes. For that, it is suggested that corticosteroids modulate the activity of the disease by suppressing the immune system.

DETAILED DESCRIPTION:
Fulminant hepatic failure (FHF) in children is a potentially devastating disease. The mortality rate may reach 80-90% in the absence of liver transplantation. FHF is the clinical manifestation of liver cell death of a critical degree with insufficient hepatocellular regeneration and characterized by coagulopathy with or without hepatic encephalopathy.

Liver injury is considered to be mainly immune mediated with augmentation of cytolytic pathways of infected hepatocytes. For that, it was suggested that corticosteroids modulate the activity of the disease by suppressing the immune system.

ELIGIBILITY:
Inclusion Criteria:

The patient is diagnosed to have FHF, if he fulfilled all the following criteria:

1. Evidence of liver dysfunction within 8 weeks of onset of symptoms (neonates may have only deranged liver functions without overt symptoms).
2. Uncorrectable coagulopathy (6-8 hours after administration of one dose of parenteral vitamin K) with International Normalized Ratio (INR) >1.5 in patients with hepatic encephalopathy, or INR> 2.0 in patients without encephalopathy.
3. No evidence of chronic liver disease.

Exclusion Criteria:

1. Presence of absolute contra-indications to steroid therapy (as presence of an active gastrointestinal bleeding, renal failure, acute pancreatitis, active tuberculosis, uncontrolled diabetes and psychosis).

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 33 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Side effect 1 Number of patients with anaphylaxis | 2 months
  Number of patients with anaphylaxis
Side effect 2 Number of patients with angioedema | 2 months
  Number of patients with angioedema
Side effect 3 Number of patients with cardiac arrest | 2 months
  Number of patients with cardiac arrest
Side effect 4 Number of patients with arrhythmias | 2 months
  Number of patients with arrhythmias
Side effect 5 Number of patients with circulatory collapse | 2 months
  Number of patients with circulatory collapse
Side effect 6 Number of patients with congestive heart failure | 2 months
  Number of patients with congestive heart failure
Side effect 7 Number of patients with pulmonary edema | 2 months
  Number of patients with pulmonary edema
Side effect 8 Number of patients with pancreatitis | 2 months
  Number of patients with pancreatitis

SECONDARY OUTCOMES:
Efficacy 1 Number of survivors | 2 months
  number of living patients
Efficacy 2 Number of deaths | 2 months
  number of died patients
Efficacy 3 serum prothrombin time | 72 hour
  serum prothrombin time
Efficacy 3 grade of encephalopathy | 72 hour
  grade of encephalopathy
Efficacy 4 duration of encephalopathy | 2 months
  duration of encephalopathy

CONTACTS AND LOCATIONS:
Overall Officials: Hanaa El-Araby, M.D., Principal Investigator — Pediatric Hepatology Department, National Liver Institute, Egypt; Mostafa M Sira, M.D., Study Director — Pediatric Hepatology Department, National Liver Institute, Egypt; Haydi M Zakaria, M.Sc., Study Chair — Quesna Central Hospital, Ministry Of Health, Egypt; Tahany A Salem, M.Sc., Study Chair — Pediatric Hepatology Department, National Liver Institute, Egypt
Locations (1):
- National Liver Institute, Menoufia, Menoufia, Egypt

REFERENCES:
- [Background] Cochran JB, Losek JD. Acute liver failure in children. Pediatr Emerg Care. 2007 Feb;23(2):129-35. doi: 10.1097/PEC.0b013e3180308f4b. PMID 17351416
- [Background] Bernal W, Auzinger G, Dhawan A, Wendon J. Acute liver failure. Lancet. 2010 Jul 17;376(9736):190-201. doi: 10.1016/S0140-6736(10)60274-7. PMID 20638564
- [Background] Fujiwara K, Kojima H, Yasui S, Okitsu K, Yonemitsu Y, Omata M, Yokosuka O. Hepatitis A viral load in relation to severity of the infection. J Med Virol. 2011 Feb;83(2):201-7. doi: 10.1002/jmv.21958. PMID 21181913
- [Background] Fujiwara K, Yasui S, Yonemitsu Y, Fukai K, Arai M, Imazeki F, Suzuki A, Suzuki H, Sadahiro T, Oda S, Yokosuka O. Efficacy of combination therapy of antiviral and immunosuppressive drugs for the treatment of severe acute exacerbation of chronic hepatitis B. J Gastroenterol. 2008;43(9):711-9. doi: 10.1007/s00535-008-2222-5. Epub 2008 Sep 20. PMID 18807133
- [Background] Lahuna O, Rastegar M, Maiter D, Thissen JP, Lemaigre FP, Rousseau GG. Involvement of STAT5 (signal transducer and activator of transcription 5) and HNF-4 (hepatocyte nuclear factor 4) in the transcriptional control of the hnf6 gene by growth hormone. Mol Endocrinol. 2000 Feb;14(2):285-94. doi: 10.1210/mend.14.2.0423. PMID 10674400
- [Background] Seshadri R, Feldman BM, Ilowite N, Cawkwell G, Pachman LM. The role of aggressive corticosteroid therapy in patients with juvenile dermatomyositis: a propensity score analysis. Arthritis Rheum. 2008 Jul 15;59(7):989-95. doi: 10.1002/art.23829. PMID 18576304

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-11): https://cdn.clinicaltrials.gov/large-docs/67/NCT02375867/Prot_SAP_001.pdf